CLINICAL TRIAL: NCT05312333
Title: Holter Monitoring of Critically-ill Childern in PICU at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Mohamed, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-03-12
Record Dates: First submitted 2022-03-13; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Critically Ill Childern in PICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically-ill childern

SUMMARY:
Holter Monitoring is a way to continuously check the electrical activity of the heart .

Continuous ECG recording show to be one of the most effective noninvasive clinical tools in the diagnosis of cardiac symptoms prognostic assessment and in the evaluation of many cardiac therapeutic intervention.

The clinical utility of ambulatory ECG lies in its ability to examine continuously a patient over an extended period of time, permitting patient ambulatory activity and facilitating the diurnal electrocardiographic examination of a patient in a changing environmental conditions (both physical and psychological) .

ELIGIBILITY:
Inclusion Criteria:

* 1- children admitted to pediatric department as in :
* Pediatric intensive care unit (PICU).
* Pediatric critical care unit (PCCU).
* Emergency room (ER). 2- Age from 1 month- 12 years. 3- Critical ill child fulfill these criteria:
* Persistent convulsions.
* Abnormal GCS
* Haemodynamic instability
* Foreign body inhalation
* Sever cardiac problem
* Irregular breathing
* DKA
* Others

Exclusion Criteria:1-Neonates 2-End-stage or those with end-organ failure . 3-Whom GCS is below 6. 4-Whom done cardiac catheterization for any purpose . 5-Previously done Holter. 6-Multiple traumatized patient.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill children are those children whom requiring, or potentially requiring, high reliance or serious consideration.
  There are variant emergent conditions may affect the child, such as airway problems which includes tonsillitis, airway obstruction which caused be foreign-body, pneumonia, asthma, and bronchitis, in addition to cardiac arrest and respiratory failure. There is also abdominal pain diarrhea, nausea, and vomiting. Child also may face seizures, poisoning sudden infant death syndrome (SIDS).
  * Having seizures; unusual movements.
  * No spontaneous development, unfit to sit or stand.
  * Less alert or drew in with clinician or parental figure; not resisting of the examination.
  * No interaction or eye-to-eye connection with individuals and the surrounding.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Abnormalities detecred in Holter monitoring of critically-ill childern | one year
  the relation between abnormalities detected in Holter and prognosis of critically-ill childern
The relation between heart rate variability and outcome ,prognosis of illness | one year
  Increased illness severity and poor outcomes ,the most common method of objectively assesing autonomic nervous system dysregulation is through measurement of heart rate variability ,which reflect the normal ,physiologic alternation in the intervals in the time between consecutive heart beats that occur when there is balance of sympathetic and parasympathetic inputs on the electrical conduction system of the heart.
Arrhythmia detected in critically-ill childern | one year
  arrhythmia detected in Holter of critically ill childern whom have any critical illness

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennedy HL. The history, science, and innovation of Holter technology. Ann Noninvasive Electrocardiol. 2006 Jan;11(1):85-94. doi: 10.1111/j.1542-474X.2006.00067.x. PMID 16472287
- [Background] Marsillio LE, Manghi T, Carroll MS, Balmert LC, Wainwright MS. Heart rate variability as a marker of recovery from critical illness in children. PLoS One. 2019 May 17;14(5):e0215930. doi: 10.1371/journal.pone.0215930. eCollection 2019. PMID 31100075
- [Background] Leteurtre S, Duhamel A, Salleron J, Grandbastien B, Lacroix J, Leclerc F; Groupe Francophone de Reanimation et d'Urgences Pediatriques (GFRUP). PELOD-2: an update of the PEdiatric logistic organ dysfunction score. Crit Care Med. 2013 Jul;41(7):1761-73. doi: 10.1097/CCM.0b013e31828a2bbd. PMID 23685639
- [Background] Rijnbeek PR, Witsenburg M, Schrama E, Hess J, Kors JA. New normal limits for the paediatric electrocardiogram. Eur Heart J. 2001 Apr;22(8):702-11. doi: 10.1053/euhj.2000.2399. PMID 11286528